CLINICAL TRIAL: NCT03621345
Title: Bilateral Ultrasound-Guided Erector Spinae Plane Block For Postoperative Analgesia in Breast Reduction Surgery: A Prospective, Randomized and Controlled Trial
Brief Title: Bilateral Ultrasound-Guided Erector Spinae Plane Block For Postoperative Analgesia in Breast Reduction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Demet Laflı Tunay, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CukurovaUniv
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain; Breast Hypertrophy
MeSH Terms: conditions — Pain, Postoperative; Gigantomastia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): The bilateral erector spine plane (ESP) block will be performed with ultrasound guided, preoperatively. Following antiseptic preparation of block site with povidone iodine, ultrasound probe will be placed 3 cm lateral to spine at T5 level. After identifying the erector spinae muscle and transverse process, the overlying skin will be infiltrated with local anesthetics and 20 mL local anesthetics (10 mL 0.5% bupivacaine + 10 mL 1% lidocaine) will be injected deep to the erector spinae muscle. The same procedure will be performed on the other side. Also, patients will receive intravenous patient controlled analgesia with morphine, and 1 g acetaminophen for supplemental analgesia if pain score raises over 5/10 on NRS and 50 mg meperidine for rescue analgesic for persistent pain.
  Interventions:
  Procedure: Ultrasound guided erector spinae plane block Other: Standard Pain Followup and Monitorization
  Interventions: Procedure: Erector spinae plane block
- sham block (Sham Comparator): A sham block will be performed while looking for intended location for ESP block placement. Skin will be infiltrated with local anesthetics but ESP block will not be performed, instead of ESP block 2 mL subcutaneous saline injection will be applied.
  Intervention: Sham block Other: Standard Pain Followup and Monitorization
  Interventions: Other: sham block

INTERVENTIONS:
Procedure: Erector spinae plane block — Ultrasound guided bilateral erector spinae plane block will be administered. An intravenous patient control analgesia device with morphine will be given to patients.
  Arms: ESP block group
Other: sham block — A sham block will be applied. Skin will be infiltrated with local anesthetics, and 2 mL subcutaneous saline injection will be applied.An intravenous patient control analgesia device with morphine will be given to patients.
  Arms: sham block

SUMMARY:
Erector spinae plane (ESP) block is a novel block developed by Forero to treat severe neuropathic pain and was firstly reported in 2016. Anatomical and radiological investigations in fresh cadavers indicate that its site of action is likely at the dorsal and ventral rami of the thoracic spinal nerves. The ESP block has a clear and simple sonoanatomy, it is easy to perform, not time consuming and generally well tolerated by the patients. So, the investigators believed that the ESP block may be an effective and safer alternative to paravertebral block, epidural analgesia and other myofascial thoracic wall blocks in breast surgery and designed a prospective, randomised, placebo-controlled trial for pain management.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II, 18-65 years of age, adult, female patients undergoing elective breast reduction surgery

Exclusion Criteria:

* Coagulopathy
* Allergy to amide-type local anesthetics
* Infection at the ESP block injection site
* Severe obesity (BMI > 35 kg/m2)
* Liver or renal deficiency
* Patients with anatomical deformities
* Recent use of analgesic drugs
* Patient refusal or inability to consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 24 hours
  Morphine consumption in Patient Controlled Analgesia device

SECONDARY OUTCOMES:
Intraoperative anesthetic consumption | During operation time
  Intraoperative total doses of remifentanil, pentothal, desflurane consumption
Extubation and recovery time | Through surgical operation completion
  Using modified aldrete score
Pain assessed by NRS | 24 hours
  Numeric rating scale (NRS) at rest and in motion will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Degree of sedation | 24 hours
  Ramsay Sedation Scale (RSS) will be used to assess degree of sedation. The RSS was designed as a test of arousability. The RSS scores sedation at six different levels, according to how arousable the patient is. The RSS defines the conscious state from a level 1: the patient is anxious, agitated or restless, through the continuum of sedation to a level 6: the patient is completely unresponsive.
Rate of opioid related side effects | 24 hours
  Opioid related side effects such as nause/vomiting, pruritis, bradycardia, hypotension will be evaluated at intervals up to 24 hours.
Supplemental and rescue analgesic requirement | 24 hours
  Total supplemental and rescue analgesic consumption
Patient satisfaction assessment | At the postoperative 24th hour
  It will be assessed with patient satisfaction scale classified as 'excellent': no pain, NRS=0; 'good': very mild pain, NRS=1-2; 'moderate': mild pain, NRS=3-4.
Bilateral shoulder mobility | Preoperative and postoperative 4th, 8th, 12th, and 24th hours
  It will be assessed with ability of shoulder abduction degree
Length of stay in hospital | Until discharge from hospital, up to 7 days postoperatively
  Duration of length of stay in hospital will be recorded
Rate of block related complications | Until discharge from hospital, up to 7 days postoperatively
  Rate of block related complications such as hematoma, nerve deficit, pneumothorax etc. will be recoded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Sariçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tunay DL, Ilginel MT, Karacaer F, Biricik E, Tabakan I, Ozmete O. Bilateral Ultrasound-Guided Erector Spinae Plane Block for Perioperative Analgesia in Breast Reduction Surgery: A Prospective Randomized and Controlled Trial. Aesthetic Plast Surg. 2023 Aug;47(4):1279-1288. doi: 10.1007/s00266-023-03315-0. Epub 2023 Mar 16. PMID 36928313